CLINICAL TRIAL: NCT04953611
Title: Quantitative Study on HRCT Phenotype of the GOLD COPD Assessment Staging
Brief Title: Quantitative Study on HRCT Phenotype of COPD
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013116
Record Dates: First submitted 2021-07-01; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary disease; chronic obstructive; Phenotype
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A in GOLD: CAT<10、mMRC 0-1、FEV1%≥50%、the frequency of acute exacerbations in the past year<2；
- Group B in GOLD: CAT≥10、mMRC≥2、FEV1%≥50%、the frequency of acute exacerbations in the past year<2
- Group C in GOLD: CAT<10、mMRC 0-1、 FEV1%<50%、the frequency of acute exacerbations in the past year≥2 or leading to hospital admission≥1
- Group D in GOLD: CAT≥10、mMRC≥2、FEV1%<50%、the frequency of acute exacerbations in the past year≥2 or leading to hospital admission≥1
- Control Group: not COPD

SUMMARY:
To explore the HRCT phenotype of the combined COPD assessment staging system

DETAILED DESCRIPTION:
HRCT can be rapidly and safely deployed has enabled COPD research to move beyond FEV1 by facilitating and amplifying clinical phenotyping measurements, providing quantitative information, and detecting significant responses to therapy even in the absence of significant FEV1 improvements.

We explore the HRCT phenotype of the combined COPD assessment staging system,and found that:

1. Airway remodeling occurs in COPD patients. CT shows varying degrees of bronchial wall thickness, area increasing and emphysema as the new GOLD classification Group A-D arising.
2. The GOLD Combined assessment staging system helps doctors choose an individualized treatment for the COPD patients

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 80 (including 40 and 80)
2. It meets the diagnostic criteria for COPD
3. No language communication barriers, or the family members who know the condition can complete the questionnaire on behalf of the patient, and the data are reliable;
4. Voluntarily agree to participate in this study

Exclusion Criteria:

1. Older than 80 or younger than 40
2. Pregnant women
3. Complicating with other lung diseases, such as asthma, pneumonia, bronchiectasis, lung abscess, interstitial lung disease, confirmed and suspected lung cancer of lung shadow, active pulmonary tuberculosis, etc
4. Previous lung surgery
5. Cognitive dysfunction
6. Unable to cooperate with lung function test.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consecutive outpatients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
The severity of emphysema | Within an average of 3 days after diagnosis of COPD
  % low attenuation area <950 HU (LAA %)
Indicator A of the severity of airway stenosis | Within an average of 3 days after diagnosis of COPD
  The inner diameter of bronchial (LD) in centimeter
Indicator B of the severity of airway stenosis | Within an average of 3 days after diagnosis of COPD
  The bronchial wall thickness in centimeter
Indicator C of the severity of airway stenosis | Within an average of 3 days after diagnosis of COPD
  Ratio of thickness and outer diameter (TDR)
Indicator D of the severity of airway stenosis | Within an average of 3 days after diagnosis of COPD
  % wall area for bronchial external diameter (WA%)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No